CLINICAL TRIAL: NCT03464162
Title: OnTrackNY With the Option of Social Network Meetings
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment failed. No sufficient interest in the study. Potential participants are not interested
Sponsor: Lisa Dixon (Other)
Responsible Party: Sponsor-Investigator, Lisa Dixon, Dr., New York State Psychiatric Institute
Organization: New York State Psychiatric Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7597
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2019-03

CONDITIONS: First Episode Psychosis; Schizophrenia
Keywords: Social Network Meetings; First Episode Psychosis; OnTrackNY
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Participants will choose if they want to receive Social Network Meetings or be in a group that does not receive Social Network Meetings. Entrance of clients into the study will be staggered with no more than approximately 5 individuals in the Social Network group and no more than 5 individuals not in the Social Network group enrolled each month. There will be a maximum of 15 participants (clients) in each group.
  For participants who choose Social Network Meetings, at least one member of their social network will participate in the study as well.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social Network Meetings Group (Experimental): This arm will receive Social Network Meetings for a 6 month period. Meetings may occur as often as 3 times a week when there is a crisis or more commonly would occur once every other week. These meetings will last between 60 and 90 minutes and will take place for however long the clients and their social networks would like within the project period. Ideally, each client and his/her Social Network would participate in 4 meetings during the 6 month period. This group would continue to receive care as usual with the addition of these meetings.
  *Final sample in this arm was N=3.
  Interventions: Behavioral: Social Network Meetings
- No Social Network Meetings Group (No Intervention): This arm will not receive the Social Network Meetings intervention. Clients in this arm will participate in the study for 6 months and receive care as usual during this time.
  *Final sample in this arm was N=1.
- Social Network Members (Other): This arm is comprised of individuals who are social network members of clients who are receiving the Social Network Meetings intervention.
  *Final sample in this arm was N=3 (social network members of arm 1).
  Interventions: Behavioral: Social Network Meetings

INTERVENTIONS:
Behavioral: Social Network Meetings — Social Network Meetings are a type of family therapy that includes clients and members of their social network.The social network may include family members, friends or anyone else that clients believe can help them move toward recovery. The meetings will focus on improving communication within the social network.
  Arms: Social Network Meetings Group; Social Network Members

SUMMARY:
Early intervention programs for psychosis help improve short-term treatment and recovery outcomes for individuals experiencing psychosis. OnTrackNY is a coordinated specialty care (CSC) program, developed to treat young adults within two years of experiencing a non-affective episode of psychosis. This project aims to expand the role of family engagement and support within the OnTrackNY model. Borrowing from the Needs Adapted and Open Dialogue models, the study team created a family therapy service that includes the client and members of his/her social network to navigate crises and assist in treatment planning. This service, Social Network Meetings, will be offered to individuals enrolled in the OnTrackNY@MHA program as an additional, voluntary, service option. The study proposes that the introduction of Social Network meetings may improve treatment and recovery outcomes.

DETAILED DESCRIPTION:
This project aims to expand the role of family engagement and support within the OnTrackNY model by offering a new service, Social Network Meetings. The study team will offer Social Network Meetings to individuals enrolled in the OnTrackNY@MHA program as an additional service option. This option will be completely voluntary and available for a 12 month period. Participant entrance into the study will be staggered with no more than approximately 5 individuals in the Social Network group and no more than 5 individuals not in the Social Network group enrolled each month. Participants will choose which group they would like to be in, if any. Data will be collected for all participants, both those participating and not participating in the Social Network Meetings upon entering the study and then once every three months and at the end of their time in the study. For all participants, the study will end after 6 months of participation.

Meetings may occur as often as 3 times a week when there is a crisis or more commonly would occur once every other week. These meetings will last between 60 and 90 minutes and will take place for however long the clients and their social networks would like within the project period.

Study aims are:

1. To determine the extent to which clients and their social networks find the Social Network meetings acceptable and beneficial.
2. To compare outcomes (family functioning, recovery) of individuals participating in Social Network meetings to those not participating.

ELIGIBILITY:
Subject Population 1: OnTrackNY MHA Client- Social Network Meeting Group (ages 16-30)

Inclusion Criteria:

* Ages 16-30
* Currently enrolled, clinically stable, English speaking clients in the OnTrackNY program at MHA Westchester determined my client roster for MHA Westchester program and clinical judgment
* Willingness to participate in Social Network meetings determined by self-report as asked by clinician
* Willingness to complete brief baseline and quarterly assessments determined by self-report as asked by clinician

Exclusion Criteria:

* Anyone who the OnTrackNY team determines is clinically unstable determined by clinician assessment
* Clients who are unwilling to participate in Social Network meetings determined by self-report

Subject Population 2: OnTrackNY MHA Client- No Social Network Meeting Group (ages 16-30)

Inclusion Criteria

* Ages 16-30
* Currently enrolled clients in the OnTrackNY program at MHA Westchester determined by MHA Westchester Client Roster for OnTrackNY

Exclusion Criteria:

* Anyone who the OnTrackNY team determines is clinically unstable determined by clinician assessment

Subject Population 3: Social Network Member (ages 18+)

Inclusion Criteria:

* Must be 18 years or older
* English speaking member of social network (i.e., biological or chosen family member/s) of a currently enrolled client in the OnTrackNY program at MHA Westchester who has agreed to participate in the study determined by client self-report
* Willingness to complete brief baseline and quarterly assessments determined by social network member self-report
* Willingness to participate in social network meetings determined by social network member self-report

Exclusion Criteria:

* Family members who the client does not want involved in the social network meetings determined by client self-report

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Change in score on the Questionnaire about the Process of Recovery (QPR) from baseline to 6 months | We will measure scores at baseline, 3 months and 6 months to determine change between these assessment points
  The QPR is a 15-item self-report survey which assesses individuals' perceptions of self and factors that are important to recovery. Items on the QPR are rated on a 5-point Likert scale and range from "disagree strongly" to "agree strongly."
Change in score on the SCORE-15 Index of Family Functioning and Change (SCORE-15) from baseline to 6 months | We will measure scores at baseline, 3 months and 6 months to determine change between these assessment points
  The SCORE-15 is a 15-item self-report survey which assesses perceptions about a family's level of intimacy and support for one another. It asks both clients and social network members to give impressions about the level of disclosure between family members, perceptions of trust, and how the family deals conflict and crisis.

SECONDARY OUTCOMES:
Brief Satisfaction Questionnaire | 6 Months
  We developed a brief 5-item survey that will ask clients and social network members about their satisfaction with the Social Network Meetings.

CONTACTS AND LOCATIONS:
Locations (1):
- MHA of Westchester, Yonkers, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kane JM, Robinson DG, Schooler NR, Mueser KT, Penn DL, Rosenheck RA, Addington J, Brunette MF, Correll CU, Estroff SE, Marcy P, Robinson J, Meyer-Kalos PS, Gottlieb JD, Glynn SM, Lynde DW, Pipes R, Kurian BT, Miller AL, Azrin ST, Goldstein AB, Severe JB, Lin H, Sint KJ, John M, Heinssen RK. Comprehensive Versus Usual Community Care for First-Episode Psychosis: 2-Year Outcomes From the NIMH RAISE Early Treatment Program. Am J Psychiatry. 2016 Apr 1;173(4):362-72. doi: 10.1176/appi.ajp.2015.15050632. Epub 2015 Oct 20. PMID 26481174
- [Background] Hamilton E, Carr A. Systematic Review of Self-Report Family Assessment Measures. Fam Process. 2016 Mar;55(1):16-30. doi: 10.1111/famp.12200. Epub 2015 Nov 19. PMID 26582601
- [Background] Neil, S. T., Kilbride, M., Pitt, L., Nothard, S., Welford, M., Sellwood, W., & Morrison, A. P. (2009). The Questionnaire about the Process of Recovery: A measurement tool developed in collaboration with service users. Psychosis: Psychological, Social and Integrative Approaches, 1(2), 145-155.